CLINICAL TRIAL: NCT03646734
Title: Guided Bone Regeneration With Particulate Versus Block Graft: Evaluation of the Two Techniques From the Point of View of the Physician and the Patient
Brief Title: Guided Bone Regeneration With Particulate Versus Block Graft
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Zekeriya Tasdemir, Principal investigator, TC Erciyes University
Other Study IDs: Zek
Record Dates: First submitted 2018-08-21; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Guided Bone Regeneration with Particulate graft: patients who had inadequate alveolar crest (crest width <4mm) and requested of dental implant placement, treated with guided bone regeration with particulate graft
- Guided Bone Regeneration with block graft: patients who had inadequate alveolar crest (crest width <4mm) and requested of dental implant placement, treated with guided bone regeration with block graft

SUMMARY:
The aim of present study was to compare two bone augmentation techniques (Guided Bone Regeneration, GBR, with autogenous block graft and GBR with particulate autograft plus xenograft) in terms of efficacy, complications, operational parameters (cost of the materials used, time for patient preparation, time for surgery, fatigue of the physician caused by surgery) tolerability by the patient and patient comfort.

DETAILED DESCRIPTION:
The aim of present study was to compare two bone augmentation techniques (Guided Bone Regeneration, GBR, with autogenous block graft and GBR with particulate autograft plus xenograft) in terms of efficacy, complications, operational parameters (cost of the materials used, time for patient preparation, time for surgery, fatigue of the physician caused by surgery) tolerability by the patient and patient comfort. 30 systemically healthy individuals with inadequate alveolar bone crest width who requested implant placement (15 Female and 15 Male) participated in this study. After an initial examination, 15 patients were assigned to GBR with block graft (GBR-BG) and 15 were assigned to GBR particulate autograft plus xenograft (GBR-AX). Bone thickness was recorded before surgery and at a post-operative 6th month. Complications as Bleeding, Hematoma, Flap dehiscence, Infection, Numbness were evaluated. Patients were requested to record pain and swelling via visual analog scale (VAS) at 3rd, 7th and 14th days after surgery. The swelling was also recorded by an experienced clinician at 3rd, 7th and 14th days after surgery. Cost, time for patient preparation, time for surgery, fatigue of the physician caused by surgery were also determined.

ELIGIBILITY:
Inclusion Criteria:

* 30 to 62 years of age
* systemically health
* no smoking
* no use of medications for previous 6 months
* no pregnancy and lactation
* no contraindications for periodontal surgery.

Exclusion Criteria:

* <30 and >62 years of age
* patients with systemic disease
* smoking habit ( current or past)
* any medication
* acute illness
* pregnancy or lactation

Ages: 30 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients admitted to the clinic with a complaint of tooth loss and inadequate alveolar crest (crest width <4mm) and requested of dental implant placement were examined. Patients with any systemic disease , smoking or alchol habits and medications did not included into the study due to avoid any possible effects on our results
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
bone gain | 6 month after surgery
  Bone gain was calculated by cone beam computerized tomography

SECONDARY OUTCOMES:
Pain | Post-operative pain was assessed at 3, 7, and 14 days.
  Pain was evaluated by visual analog scale Visual analog scale (VAS) consist of 10 units, in combination with a graphic rating scale. On the VAS, the left and right end of the graphic represented the absence of pain (score 0) and the most severe pain (score 10), respectively. Patients were warned to fulfill the VAS, taking into consideration the intensity of their pain in the previous 24 hours on all recall days.

CONTACTS AND LOCATIONS:
Overall Officials: Zekeriya Taşdemir, Phd, Principal Investigator — TC Erciyes University

IPD SHARING:
Plan to Share IPD: Undecided